CLINICAL TRIAL: NCT05253599
Title: Effect of Different Exercise Training Methods on the Radiographic and Inflammatory Biomarkers (CRP, TNF-α, IL-2, IL-4, IL-6) in Chronic Low Back Pain: A Randomized Control Study.
Brief Title: Radiographic and Inflammatory Biomarker Changes in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Associate Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RHPT/019/036
Record Dates: First submitted 2022-01-31; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Low Back Pain
Keywords: Isokinetic training; Virtual reality training; Cross sectional area; muscle thickness; inflammatory biomarkers; chronic low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study was a double-blinded randomized control study and the subjects were randomized and allocated equally according to the computer random table method in a 1:1:1 ratio in three groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the design and settings of the study, it was not possible to blind the treating therapist involved in the study. The subject and the therapist who was assessing the outcomes at baseline and after 4 weeks were blinded. Hence, the treating and assessing therapists were different persons and the assessing therapist remains blinded to the subject's treatment group. Subjects were instructed not to disclose their study procedures and treatment protocol with fellow-subjects and the assessing therapist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isokinetic training (Experimental): In the IKT group before isokinetic training, the subjects were asked to perform five minutes' warm-up followed by slow stretching of back extensors and flexors. The subject was asked to be in an isokinetic dynamometer (Biodex Corporation, New York, USA) in a vertical standing position.
  Interventions: Device: Isokinetic training
- Virtual reality training (Experimental): The VRT group received virtual reality training with (Pro-Kin system PK 252 N Techno body, Pelvic Module balance trunk MF, Italy) focusing on the balance of core stability muscles.
  Interventions: Device: Virtual reality training
- Control group (Active Comparator): The Control group focused on conventional balance training for core muscles. The training includes active isotonic and isometric exercise for abdominal muscles (Internal oblique, external oblique, transverse abdominus and Rectus abdominus) deep abdominal muscles (Psoas major, Psoas minor, Illiacus and Quadratus Lumborum) and back muscles (Erector spinae, Transverses spinalis, inter spinalis and Inter transverse).
  Interventions: Other: Exercises

INTERVENTIONS:
Device: Isokinetic training — The knees were flexed slightly at 15 degrees, and the fixation straps were tied around the popliteus, thigh, pelvis, chest and scapula to prevent the tricky movements.
  Arms: Isokinetic training
Device: Virtual reality training — Training was given in the sitting position which provides challenges to the balance activities of the participant. The game which was used in the current study was a shooting game, which consists of the subject sitting on the virtual platform and visualizing the game on the display screen. The game was executed and controlled by moving the trunk back and forth and left and right according to the signs. Participants can perform all the six movements of their spine within their pain limits.
  The level of difficulty of the exercises was increased by graded activity, in which the activities were gradually getting difficult and harder as participants required more muscle activity and movement.
  Arms: Virtual reality training
Other: Exercises — They performed these exercises 10-15 reps/day for 5 days per week for 4 weeks. Stretching was focused on each muscle group for 3 repetitions for 10 seconds per muscle group (Hamstring, Hip flexors and Lumbar Extensors).7 A home-based exercise protocol was prescribed to all the subjects to perform at home. All the subjects in three groups were undergone hot pack therapy for 20 mins and ultrasound with a frequency of 1 Mhz and intensity of 1.5 W/cm2 in continuous form for five minutes.
  Arms: Control group

SUMMARY:
OBJECTIVE: To find and compare the effects of isokinetic training and virtual reality training on pain intensity, trunk muscle strength, radiographical (muscle cross-sectional area and muscle thickness), and biochemical effects in chronic low back pain (LBP) patients.

DETAILED DESCRIPTION:
OBJECTIVE: To find and compare the effects of isokinetic training and virtual reality training on pain intensity, trunk muscle strength, radiographical (muscle cross-sectional area and muscle thickness), and biochemical effects in chronic low back pain (LBP) patients.

METHODS: Randomized, double-blinded controlled study was conducted on 60 LBP patients and they were divided into isokinetic training (IKT; n=20), virtual reality training (VRT; n=20), and a control group (n=20). The VRT group received virtual training for core muscles of the trunk, the IKT group received training for trunk muscles through an Isokinetic dynamometer and the control group received conventional trunk balance exercises. Pain intensity (visual analog scale -VAS), trunk muscle strength, radiographical (muscle cross-sectional area through Magnetic resonance imaging - MRI & muscle thickness through Ultrasound - US), and biochemical (CRP, TNF-α, IL-2, IL-4, IL-6) variables were measured at baseline and after 4 weeks (short term effect) of training.

ELIGIBILITY:
Inclusion Criteria:

* University male football players
* Age group of 18 - 25 years
* chronic (≥3 months) LBP,
* 4 to 8 pain intensity in visual analog scale (VAS).

Exclusion Criteria:

* Participants with severe musculoskeletal, neural, somatic, and psychiatric conditions,
* Waiting for spine surgery,
* Having alcohol or drug abuse,
* Involved in other weight and balance training programs.
* Participants with other soft tissue injuries, fractures in the lower limbs and pelvic bone, deformities.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — University male football players in the age group of 18 - 25 years
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | At Baseline
  The pain intensity was measured by visual analog scale (VAS) which consist of a 10 cm horizontal line representing one end with "no pain at all" and the other end with "as bad as possible it could be." Each subject was asked to enter in the line as per his pain perception at rest and the score was measured by the distance on the line. The reliability and validity of VAS in application of musculoskeletal conditions was good.
Pain Intensity | After 4 weeks
  The pain intensity was measured by visual analog scale (VAS) which consist of a 10 cm horizontal line representing one end with "no pain at all" and the other end with "as bad as possible it could be." Each subject was asked to enter in the line as per his pain perception at rest and the score was measured by the distance on the line. The reliability and validity of VAS in application of musculoskeletal conditions was good.
Trunk flexor & extensor muscle strength | At Baseline
  The trunk flexor and extensor muscles' peak torque was measured by using isokinetic dynamometer. The participant was positioned in standing position and wrapped the lower extremities with Velcro straps to prevent trick movements. Three measurements were taken at 900 per second for trunk flexors and extensors and the average value was considered for data analysis. The reliability and validity of this method of application in low back pain condition was good.
Trunk flexor & extensor muscle strength | After 4 weeks
  The trunk flexor and extensor muscles' peak torque was measured by using isokinetic dynamometer. The participant was positioned in standing position and wrapped the lower extremities with Velcro straps to prevent trick movements. Three measurements were taken at 900 per second for trunk flexors and extensors and the average value was considered for data analysis. The reliability and validity of this method of application in low back pain condition was good.

SECONDARY OUTCOMES:
Para spinal CSA | Baseline and after 4 weeks
  Cross sectional area (CSA) is an area exposed by cut through at right angles to an axis. T2 weighted images of para spinal muscles (PM: Psoas Major, QL: Quadratus Lumborum, Mf: Multifidus and ES: Erector Spinae) CSA were taken using a 3-T MRI-scanner (Closed MRI system, Siemens, Hamburg, Germany) with a slice thickness of 5 mm. The subjects were placed in a supine position with a pillow kept under the knees to maintain the normal lordosis of the lumbar spine. The CSA at the level of L3-L4 was selected because of their maximal size at this level.
Muscle thickness | Baseline and after 4 weeks
  Muscle size is considered as the thickness of muscle and the thickness of Multifidus muscle was measured by the diagnostic ultrasound device (Hitachi Ultrasound, Tokyo, Japan) which is the most reliable and valid method of measurement. The thickness of multifidus was taken from the left and right side of the L4 and L5 level. The subject lies in a prone position with a pillow under the abdomen to maintain lordosis. The thickness of the muscle was measured by measuring the distance between the most superficial portion of the facet joint and the plane between the muscle and the skin.
Inflammatory Biomarker | Baseline and after 4 weeks
  Subject's blood samples of 10 ml were taken in sterile tubes between 08:00 - 10:00 am. Serum was separated and centrifuged, which was frozen at -700 C and stored. Serum levels of CRP, TNF-α, IL-2, IL-4, IL-6 were measured by enzyme-linked immunosorbent assay (ELISA) technique. The kit was used according to the guidelines of the manufacturer. The lower and upper limits of detection were computed for each assay, and the average percentages of samples were reported for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data can be obtained by contacting the principal investigator
Supporting Information: Study Protocol, ICF
Time Frame: 4 weeks